CLINICAL TRIAL: NCT00996697
Title: A Proof Of Concept Study To Evaluate Tiotropium as Add-on Therapy to Inhaled Budesonide/Formoterol Combination in COPD
Brief Title: Differential Trough Effects of 'Triple Therapy' on Pulmonary Function in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: FARD12
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FARD12
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: COPD
Keywords: COPD (chronic obstructive pulmonary disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triple therapy (Active Comparator): Symbicort and tiotropium
  Interventions: Drug: Budesonide/formoterol and tiotropium
- Combination therapy (Placebo Comparator): Symbicort and placebo
  Interventions: Drug: Budesonide/formoterol and placebo

INTERVENTIONS:
Drug: Budesonide/formoterol and tiotropium — Symbicort 200/2, 2puff bid plus tiotropium 18mcg/day
  Arms: Triple therapy
Drug: Budesonide/formoterol and placebo — Symbicort 200/6 2puff bid and placebo
  Arms: Combination therapy

SUMMARY:
Different medications are often used in combination for the condition COPD (chronic obstructive pulmonary disease). Some medicines act by opening the airways (bronchodilators) and some act as anti-inflammatories (steroids). More recently an approach of using a combination inhaler (containing a steroid and a long-acting bronchodilator) at the same time as a long acting bronchodilator of a different group of medicines (anti-cholinergics inhalers) has been used. This approach is sometimes called 'triple therapy'. Studies which have looked at these combinations usually use only standard blowing tests (spirometry) to test these medicines and focus on the effects of the medicines at their highest (peak) levels. It is some ways more relevant to study these medicines towards to end of the dose period (trough)- just before the next dose. This is when there is less medicine in the system, and differences in drug effects are more obvious. There are also more detailed breathing tests than spirometry which get a more detailed picture of the way the lungs respond to bronchodilator medicines. The investigators have studied 'triple therapy' in COPD, by measuring the effects at the end of the dosing interval (trough) using a range of detailed respiratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Current or ex-smokers
* aged over 50years
* FEV1/FVC ratio less than 0.7
* FEV1 less than 60% predicted

Exclusion Criteria:

* Diagnosis of asthma, ABPA or bronchiectasis
* Recent RTI or steroid use
* Inability to perform study procedures or to give informed consent
* Known sensitivity to trial medications

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in trough FEV1 for tiotropium compared to placebo when added to formoterol/budesonide combination | 2 weeks

SECONDARY OUTCOMES:
Change in IOS and bodyplethysmography at trough for tiotropium compared to placebo when added to formoterol/budesonide combination | 2 weeks
Change in spirometry, IOS and Bodyplethysmography at trough for formoterol/budesonide compared to washed-out baseline | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma and Allergy Research Group, Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Result] Williamson PA, Short PM, Clearie KL, Vaidyanathan S, Fardon TC, Howaniec LJ, Lipworth BJ. Paradoxical trough effects of triple therapy with budesonide/formoterol and tiotropium bromide on pulmonary function outcomes in COPD. Chest. 2010 Sep;138(3):595-604. doi: 10.1378/chest.10-0247. Epub 2010 Apr 23. PMID 20418370